CLINICAL TRIAL: NCT02952898
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Comparison Study to Determine the Therapeutic Equivalence of GDC 695 and Diclofenac Sodium Gel, 3% in Subjects With Actinic Keratoses
Brief Title: Study Comparing GDC 695 and Diclofenac Sodium Gel, 3% in Subjects With Actinic Keratoses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Balmoral Medical company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDC-695-001
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Results first posted 2019-01-10 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Actinic Keratosis
Keywords: solar keratoses
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Drug (Experimental): GDC 695 gel applied topically as directed.
  Interventions: Drug: GDC 695
- Reference Drug (Active Comparator): Diclofenac sodium gel, 3% applied topically as directed.
  Interventions: Drug: Diclofenac Sodium Gel, 3%
- Placebo (Placebo Comparator): Vehicle gel applied topically as directed.
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: GDC 695 — GDC 695 is a topical gel.
  Arms: Test Drug
Drug: Diclofenac Sodium Gel, 3% — Diclofenac sodium gel, 3% is an FDA-approved drug.
  Arms: Reference Drug
Drug: Vehicle gel — Vehicle topical gel contains 0.0% of active drug and is color matched to the other two active test drugs.
  Arms: Placebo

SUMMARY:
This research study is being done to compare the safety and effectiveness of GDC 695 (test drug) against the currently marketed reference drug (diclofenac sodium gel, 3%) and to establish that these two drugs work better than placebo in the treatment of actinic keratosis.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent.
* Immunocompetent male and/or non-pregnant female, 18 years of age or older.
* Willing and able to apply the test article(s) as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
* Clinical diagnosis of actinic keratosis.
* In good general health and free of any disease state or physical condition.
* Women, must be post-menopausal, surgically sterile, or use an effective method of birth control with a negative urine pregnancy test (UPT) at the Baseline Visit (Day 1).

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or are planning to become pregnant or breastfeed during the study.
* Is currently enrolled in another investigational drug or device study or has used an investigational drug or investigational device within 30 days prior to the Baseline Visit (Day 1).
* Has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the study.
* Is immunosuppressed (e.g., human immunodeficiency virus [ HIV], systemic malignancy, graft host disease, etc.) or is taking medications that suppress the immune system.
* Has experienced an unsuccessful outcome from previous topical diclofenac sodium therapy.
* Has a history of sensitivity to any of the ingredients in the test articles or other excipients in the test or reference drug.
* Has signs or symptoms consistent with the aspirin (ASA) triad.
* Has used topical medications: corticosteroids, alpha hydroxy acids (e.g., glycolic acid, lactic acid, etc. >5%), beta hydroxy acid (salicylic acid >2%), urea >2%, 5-fluorouracil, diclofenac, imiquimod, ingenol mebutate, aminolevulinic acid (ALA) or prescription retinoids (e.g., tazarotene, adapalene, tretinoin), over-the-counter (OTC) products labeled as scrubs of any kind which are used to smooth the skin (as they contain some form of exfoliant such as nut shells, coffee grounds, polymer particles, etc.) within the selected treatment area (face or bald scalp) within one month prior to the Baseline Visit.
* Has had cryodestruction or chemodestruction, curettage, photodynamic therapy (PDT), surgical excision, or other treatments for AK within the selected treatment area (face or bald scalp) within one month prior to the Baseline Visit.
* Has used oral corticosteroid therapy, interferon, cytotoxic drugs, immunomodulators, immunosuppressive therapies, or retinoids within one month prior to the Baseline Visit.
* Has used oral isotretinoin within six months prior to the Baseline Visit.
* Has used chemical peels, including but not limited to alphahydroxy acid, betahydroxy acid, bichloroacetic acid, trichloroacetic acid, and phenol within the selected treatment area (face or bald scalp) within six months prior to the Baseline Visit.
* Has had dermatologic procedures or surgeries such as: laser resurfacing, PUVA (Psoralen + ultraviolet A) therapy, ultraviolet B (UVB) therapy, ALA-PDT, or dermabrasion within the selected treatment area (face or bald scalp) within six months prior to the Baseline Visit.
* Has lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the selected treatment area (face or bald scalp).
* Has active gastrointestinal ulceration or bleeding or has a history of gastrointestinal bleeds due to use of aspirin or other NSAIDs.
* Has severe renal or hepatic impairment.
* Has any condition which, in the investigator's opinion, could interfere with the evaluation of the test drugs or that could make it unsafe or preclude the subject's ability to fully participate in this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Site 07, Fort Smith, Arkansas
  - Site 14, San Diego, California
  - Site 24, San Ramon, California
  - Site 22, Clearwater, Florida
  - Site 01, North Miami Beach, Florida
  - Site 27, Ocala, Florida
  - Site 12, Tampa, Florida
  - Site 05, Carmel, Indiana
  - Site 02, Plainfield, Indiana
  - Site 25, Saint Joseph, Missouri
  - Site 21, Albuquerque, New Mexico
  - Site 03, Warwick, Rhode Island
  - Site 26, Anderson, South Carolina
  - Site 04, Greenville, South Carolina
  - Site 28, Norfolk, Virginia
  - Site 10, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 2016 to July 2017
  The location of clinical sites included dermatology clinics and clinical research centers.
Pre-assignment Details: All subjects who met the entry criteria and were randomized and enrolled into the study.
Groups:
- GDC 695 Gel: The test drug is GDC 695 gel applied topically as directed.
  GDC 695: GDC 695 is a topical gel.
- Diclofenac Sodium Gel: The reference drug is Diclofenac sodium gel, 3% applied topically as directed.
  Diclofenac Sodium Gel, 3%: Diclofenac sodium gel, 3% is an FDA-approved drug.
Period: Overall Study
Arm/Group | GDC 695 Gel | Diclofenac Sodium Gel | Placebo
Started | 220 | 221 | 224
Completed | 198 | 202 | 209
Not Completed | 22 | 19 | 15
Not completed — Withdrawal by Subject | 10 | 8 | 8
Not completed — Adverse Event | 8 | 8 | 3
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — Non-compliance with study drug | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline demographic information is based on the safety population, which includes all randomized subjects who received at least one dose of the test article. Four subjects (2 in Test Drug group, 1 in Reference Drug group, and 1 in Placebo group) were excluded for not applying any test article.
Groups:
- GDC 695 Gel: GDC 695 gel applied topically as directed.
  GDC 695: GDC 695 is a topical gel.
- Diclofenac Sodium Gel: Diclofenac sodium gel, 3% applied topically as directed.
  Diclofenac Sodium Gel, 3%: Diclofenac sodium gel, 3% is an FDA-approved drug.
- Total: Total of all reporting groups
Arm/Group | GDC 695 Gel | Diclofenac Sodium Gel | Placebo | Total
Number analyzed (Participants) | 218 | 220 | 223 | 661
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (9.4) | 69.6 (9.8) | 69.1 (9.3) | 69.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 45 | 36 | 112
  Male | 187 | 175 | 187 | 549
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 14 | 13 | 16 | 43
  Ethnicity: Not Hispanic or Latino | 204 | 207 | 207 | 618
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 2 | 1 | 4
  Race: White | 217 | 218 | 222 | 657
Region of Enrollment [Number; unit: participants]
  United States | 218 | 220 | 223 | 661

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Complete Clearance of AK Lesions
Description: Complete Clearance was defined as 100% clearance of all Actinic Keratosis (AK) lesions (having a count of zero AKs) in the treatment area (face or bald scalp) at the Day 90 visit (30 Days Post Treatment).
Time Frame: Day 90 (30 days after completion of 60 days of treatment)
Population: Analysis shown is based on the modified Intent-to-Treat (mITT) population, defined as all randomized subjects who met the following requirements, 1) met all inclusion/exclusion criteria; 2) applied at least one dose of test article; 3) and returned for at least one post-baseline evaluation clinic visit (Visits 3, 5, or 6).
Measure: Number; unit: percentage of participants
Arm/Group | GDC 695 Gel | Diclofenac Sodium Gel | Placebo
Number analyzed (Participants) | 215 | 218 | 221
percentage of participants | 30.2 | 25.7 | 9.5
Statistical Analysis 1: Comparison: GDC 695 Gel vs Placebo; Two-sided, continuity-corrected Chi-square tests was used to evaluate the superiority of GDC 695 gel's complete clearance proportion over that of the Vehicle treatment in the mITT population using LOCF; Test type: Superiority; p < 0.0001, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Diclofenac Sodium Gel vs Placebo; Two-sided, continuity-corrected Chi-square tests was used to evaluate the superiority of Diclofenac sodium gel's complete clearance proportion over that of the Vehicle treatment in the mITT population using LOCF; Test type: Superiority; p < 0.0001, Chi-squared, Corrected

2. Other Pre Specified Outcome: Adverse Events (AEs)
Description: AEs will be assessed by the investigator and the incidence (severity and causality) of any local and systemic AEs will be reported.
Time Frame: Day 0 through Day 90
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) were collected from study Day 1 (enrollment/first dose) to study completion (Day 90) or participant termination. AEs that continued beyond completion/termination were followed until resolution or stabilization.
Description: There were a total of four (4) Serious Adverse Events (SAEs) in three (3) subjects in the Reference group (Diclofenac sodium gel); one of these subjects experienced two (2) SAEs: (1) Bladder transitional cell carcinoma and (2) Haematuria. There were a total of six (6) SAEs in the five (5) subjects in the Placebo group (Vehicle gel); one of these subjects experienced two (2) SAEs: (1) Flank pain and (2) Lung infiltration.
Groups:
- GDC 695: GDC 695 gel applied topically as directed.
  GDC 695: GDC 695 is a topical gel.
Arm/Group | GDC 695 | Diclofenac Sodium Gel | Placebo
All-Cause Mortality (participants affected / at risk) | 0/218 | 0/220 | 0/223
Serious Adverse Events (participants affected / at risk) | 1/218 | 3/220 | 5/223
Other Adverse Events (participants affected / at risk) | 19/218 | 14/220 | 6/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC 695 (N=218) | Diclofenac Sodium Gel (N=220) | Placebo (N=223)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC 695 (N=218) | Diclofenac Sodium Gel (N=220) | Placebo (N=223)
Application site erythema (General disorders) | 4 (4) | 3 (3) | 1 (1)
Application site oedema (General disorders) | 3 (3) | 2 (2) | 0 (0)
Application site pain (General disorders) | 3 (3) | 1 (1) | 1 (1)
Application site pruritus (General disorders) | 3 (3) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Investigator, including all employees and coworkers involved with this study, agree not to publish the results of this study without the prior written consent of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT02952898/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT02952898/SAP_001.pdf